CLINICAL TRIAL: NCT04634058
Title: PD-L1 Antibody Combined With CTLA-4 Antibody for Patients With Advanced Intrahepatic Cholangiocarcinoma Who Progressed After Standard Treatment: a Single-arm, Phase II Clinical Study
Brief Title: PD-L1 Antibody Combined With CTLA-4 Antibody for Patients With Advanced Intrahepatic Cholangiocarcinoma Who Progressed After Standard Treatment
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: zs-ICC-PDCT
Record Dates: First submitted 2020-11-17; First posted 2020-11-18 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Cholangiocarcinoma, Intrahepatic; PD-L1; CTLA4
MeSH Terms: conditions — Cholangiocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- PD-L1 antibody combined with CTLA-4 antibody (Experimental): After 4 cycles of PD-L1 antibody combined with CTLA-4 antibody treatment, PD-L1 monotherapy was maintained until the disease progressed or intolerable toxicity and adverse reactions or the medication was used for two years.
  Interventions: Drug: PD-L1 antibody combined with CTLA-4 antibody

INTERVENTIONS:
Drug: PD-L1 antibody combined with CTLA-4 antibody — After 4 cycles of PD-L1 monoclonal antibody combined with CTLA-4 monoclonal antibody treatment, PD-L1 monotherapy was maintained until the disease progressed or intolerable toxicity and adverse reactions or the medication was used for two years.

SUMMARY:
The study aims to evaluate the efficacy and safety of PD-L1 antibody combined with the CTLA-4 antibody in patients with advanced ICC who progressed after standard treatment.

DETAILED DESCRIPTION:
The prognosis of unresectable and metastatic intrahepatic biliary tract cancer (ICC) is extremely poor. The median overall survival of first-line gemcitabine and cisplatin for advanced biliary tumors (including ICC) is only 11.7 months. Currently, there is no standard second-line or third-line treatment for advanced ICC, and there is an urgent need to develop new treatment methods to improve patient survival. Chronic inflammation caused by viral infections and bile duct stones is the most common potential risk factor for ICC. The abnormal immune system plays a key role in the occurrence and development of ICC. The immune checkpoint molecules PD-L1 and CTLA-4 are overexpressed in ICC, and they are obviously heterogeneous, so immunotherapy has potential value. Immune checkpoint inhibitors against PD-1/PD-L1 show a good objective remission rate in advanced biliary tumors (including ICC). CTLA-4 inhibitors combined with PD-1/PD-L1 inhibitors show significant clinical enhancement Role, CTLA-4 inhibitors combined with PD-1/PD-L1 inhibitors have been clinically studied in a number of solid tumors. In this phase II clinical study, we will evaluate the efficacy and safety of PD-L1 monoclonal antibody combined with CTLA-4 monoclonal antibody in patients with advanced ICC who progressed after standard treatment.

ELIGIBILITY:
Inclusion Criteria:

1. For unresectable or metastatic or postoperative recurrence, histologically confirmed advanced ICC, provide enough tissue samples for PD-L1, CTLA-4 immunohistochemistry, and exome sequencing
2. The standard systemic treatment of advanced ICC (gemcitabine or platinum or fluorouracil) failed due to disease progression or toxicity
3. There are measurable lesions defined by RECIST standard v1.1
4. For patients with a history of liver chemoembolization, radiofrequency ablation/intervention, or radiotherapy, there must be measurable lesions outside the chemoembolization or radiotherapy area or measurable progression lesions at the chemoembolization or radiotherapy site
5. ECOG physical strength status ≤ 1
6. Life expectancy> 3 months
7. Adequate renal function: creatinine (Cr) ≤ 1.5 × upper limit of normal (ULN) or glomerular filtration rate (GFR) ≥ 60mL/min/1.73 m2
8. Sufficient liver function: bilirubin ≤ 1.5 × ULN and alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 5 × ULN
9. Sufficient bone marrow reserve: absolute value of neutrophils (ANC)> 1500/mcl, platelets (Plts)> 75,000/mcl, hemoglobin (Hgb) ≥ 9.0g/dl
10. Prothrombin time/activated partial thromboplastin time (PT/PTT) <1.5 × ULN
11. Age ≥18 years old
12. HBV infected persons must meet the following criteria to be eligible to participate in the study:

    Chronic hepatitis B virus (HBV) infection (defined as hepatitis B surface antigen [HBsAg] positive and/or detectable HBV DNA) subjects must have HBV viral load below 2000 IU/ml before the first dose of the study intervention. Active HBV-treated subjects with a viral load of less than 2000 IU/ml should receive antiviral therapy throughout the study intervention period and check the HBV viral load every 6 weeks. Subjects whose HBV infection is clinically cured (defined as HBsAg negative and anti-HBc positive) and whose HBV viral load cannot be detected during screening should be checked for HBV viral load every 6 weeks. If the viral load exceeds 2000 IU/ml, HBV treatment should be carried out. Antiviral treatment after completing the research intervention should follow local guidelines.
13. The toxicity of the previous treatment has been restored to ≤1 grade (if there is surgery, the wound has completely healed)
14. Female subjects of childbearing age must undergo a pregnancy test within 2 weeks before starting the study medication, and the result is negative, and are willing to use a medically approved high-efficiency contraceptive method during the study period and within 24 weeks after the last study drug administration (Such as intrauterine device, contraceptive pills or condoms); for male subjects whose partners are females of childbearing age, they should agree to use effective methods of contraception during the study period and within 24 weeks after the last study administration
15. Subjects voluntarily joined the study, signed an informed consent form, had good compliance, and cooperated with follow-up.

Exclusion Criteria:

1. Past treatment with CTLA-4 mAb
2. Hilar cholangiocarcinoma or extrahepatic cholangiocarcinoma or periampullary carcinoma or gallbladder cancer
3. Major surgery or radiotherapy within 4 weeks before enrollment
4. Active, known, or suspected autoimmune diseases
5. Congestive heart failure or symptomatic coronary artery disease within 3 months before enrollment
6. Cerebrovascular accident occurred in the past 6 months
7. Clinically significant bleeding, bleeding event, or thromboembolic disease occurred within 6 months
8. History of bowel perforation
9. A history of (non-infectious) pneumonia requiring steroid treatment or current pneumonia
10. Known history of human immunodeficiency virus (HIV) infection
11. History of severely impaired lung function or interstitial lung disease
12. Diagnosed concurrent malignant tumors in the past 5 years (except for fully treated non-melanoma skin cancer, superficial transitional cell carcinoma of the bladder and cervical carcinoma in situ [CIS]) or any currently active malignant tumors
13. HCV RNA positive test indicates the active period
14. Patients who have previously received allogeneic bone marrow transplantation or solid organ transplantation
15. Uncontrollable or symptomatic hypercalcemia
16. Known uncontrollable or symptomatic active central nervous system (CNS) metastasis
17. Symptomatic advanced patients who are at risk of life-threatening complications in the short term (including patients with uncontrollable large amounts of exudate [thoracic cavity, pericardium, abdominal cavity])
18. Known allergies to study drugs or excipients or known severe allergic reactions to any monoclonal antibody
19. Severe infections during screening, including but not limited to infectious complications requiring hospitalization, bacteremia, severe pneumonia, etc.
20. Have received any other experimental drug treatment or participated in another interventional clinical study within 4 weeks before signing the ICF
21. Live attenuated vaccine within 4 weeks before enrollment or planned during the study period and 60 days after the end of study drug treatment
22. Known mental illness, alcohol abuse, inability to quit smoking, drug or drug abuse, etc.
23. Past or current evidence indicates that any conditions, treatments, or laboratory abnormalities that may confuse the research results, interfere with the subject's participation in the entire research process, or the researcher believes that participating in this research is not in the subjects' best interests.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-03-26 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
objective response rate (ORR) | 12 months
  the objective response rate (ORR) of advanced ICC patients who progressed after standard treatment with PD-L1 antibody SHR-1316 combined with CTLA-4 antibody IBI310

SECONDARY OUTCOMES:
Safety: the potential side effects | 12 months
  the potiential side effects
overall survival | 18 months
  From the beginning date of combined therapy to the date of death
Progression free survival | 12 months
  From the beginning date of combined therapy to disease progresion or death, whichever occurs first

CONTACTS AND LOCATIONS:
Overall Officials: Fan Jia, MD & PhD, Principal Investigator — Shanghai Zhongshan Hospital
Locations (1):
- Zhongshan hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lu JC, Zeng HY, Sun QM, Meng QN, Huang XY, Zhang PF, Yang X, Peng R, Gao C, Wei CY, Shen YH, Cai JB, Dong RZ, Shi YH, Sun HC, Shi YG, Zhou J, Fan J, Ke AW, Yang LX, Shi GM. Distinct PD-L1/PD1 Profiles and Clinical Implications in Intrahepatic Cholangiocarcinoma Patients with Different Risk Factors. Theranostics. 2019 Jul 9;9(16):4678-4687. doi: 10.7150/thno.36276. eCollection 2019. PMID 31367249
- [Background] Lim YJ, Koh J, Kim K, Chie EK, Kim S, Lee KB, Jang JY, Kim SW, Oh DY, Bang YJ. Clinical Implications of Cytotoxic T Lymphocyte Antigen-4 Expression on Tumor Cells and Tumor-Infiltrating Lymphocytes in Extrahepatic Bile Duct Cancer Patients Undergoing Surgery Plus Adjuvant Chemoradiotherapy. Target Oncol. 2017 Apr;12(2):211-218. doi: 10.1007/s11523-016-0474-1. PMID 28084572